CLINICAL TRIAL: NCT00240500
Title: Long-Term Follow Up Study at Years 16-20, to Evaluate the Persistence of Immune Response of GlaxoSmithKline Biologicals' Hepatitis B Vaccine in Newborns of HBeAg+ and HBsAg+ Mothers
Brief Title: Follow-up Study 16-20 Years After Primary Vaccination Against Hepatitis B of Newborns From HBeAg+ & HBsAg+ Mothers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100448
Record Dates: First submitted 2005-10-13; First posted 2005-10-18 (Estimated); Results first posted 2009-05-01 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B
Keywords: Long-term follow-up; Hepatitis B antibody persistence
MeSH Terms: conditions — Hepatitis B

ARMS (6):
- HBV-1 Group (Experimental): neonates born to HBsAg+ and HBeAg+ mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
  Interventions: Biological: Engerix™-B
- HBV-2 Group (Experimental): neonates born to HBsAg+ and HBeAg+ mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
  Interventions: Biological: Engerix™-B
- HBV-3 Group (Experimental): neonates born to HBsAg+ and HBeAg- mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
  Interventions: Biological: Engerix™-B
- HBV-4 Group (Experimental): neonates born to HBsAg+ and HBeAg- mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
  Interventions: Biological: Engerix™-B
- HBV-5 Group (Experimental): neonates born to HBsAg- and HBeAg- mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
  Interventions: Biological: Engerix™-B
- HBV-6 Group (Experimental): neonates born to HBsAg- and HBeAg- mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Engerix™-B — In the primary study, subjects received HBV (10 milligram) vaccine according to a 0, 1 and 2 month schedule with a booster dose at Month 12. Subjects in the 5-dose vaccination regimen received a booster dose of HBV vaccine at Month 60.

SUMMARY:
The purpose of this study is to evaluate the persistence of anti-hepatitis B surface antigen (anti-HBs) antibodies 16, 17, 18, 19 and 20 years after administration of the first dose of the study vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The primary study was designed to evaluate the immunogenicity and protective efficacy of hepatitis B vaccine in newborns of HBeAg+ and HBsAg+ mothers in comparison with a historical control group.

The present study is carried out to evaluate the anti-HBs persistence 16-20 years after the first vaccine dose and to further investigate the prevalence and incidence of other hepatitis B markers and the clinical significance of these at all time points from Year 16-20.

No additional subjects will be recruited during this long-term follow-up study and no vaccine will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had received at least one dose of the study vaccine in the primary study (103860/064)
* Written informed consent obtained from each subject before each blood sampling visit

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2003-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Leroux-Roels G, Kuriyakose S, Leyssen M, Jacquet JM. Evidence of protection against clinical and chronic hepatitis B infection 20 years after infant vaccination in a high endemicity region. J Viral Hepat. 2011 May;18(5):369-75. doi: 10.1111/j.1365-2893.2010.01312.x. PMID 20384962
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Bock HL, Leyssen M, Jacquet JM. Persistence of antibodies and immune memory to hepatitis B vaccine 20 years after infant vaccination in Thailand. Vaccine. 2010 Jan 8;28(3):730-6. doi: 10.1016/j.vaccine.2009.10.074. Epub 2009 Nov 3. PMID 19892043
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 100448 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100448 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100448 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100448 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100448 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- HBV 5 Group: neonates born to Hepatitis B surface antigen negative (HBsAg-) and Hepatitis B e antigen negative (HBeAg-) mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
- HBV 2 Group: neonates born to Hepatitis B surface antigen positive (HBsAg+) and Hepatitis B e antigen positive (HBeAg+) mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
- HBV 1 Group: neonates born to HBsAg+ and HBeAg+ mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
- HBV 4 Group: neonates born to HBsAg+ and HBeAg- mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
- HBV 3 Group: neonates born to HBsAg+ and HBeAg- mothers who received a 5-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12 and again a booster dose at Month 60)
- HBV 6 Group: neonates born to HBsAg- and HBeAg- mothers who received a 4-dose vaccination regimen (0, 1 and 2-month schedule with a booster dose at Month 12)
Period: Overall Study
Arm/Group | HBV 5 Group | HBV 2 Group | HBV 1 Group | HBV 4 Group | HBV 3 Group | HBV 6 Group
Started | 17 | 20 | 17 | 23 | 29 | 3
Completed | 16 | 17 | 14 | 19 | 26 | 2
Not Completed | 1 | 3 | 3 | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBV 5 Group | HBV 2 Group | HBV 1 Group | HBV 4 Group | HBV 3 Group | HBV 6 Group | Total
Number analyzed (Participants) | 17 | 20 | 17 | 23 | 29 | 3 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (0.51) | 16.6 (0.5) | 16.5 (0.51) | 16.4 (0.51) | 16.8 (0.44) | 16.7 (0.58) | 16.6 (0.50)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 9 | 11 | 7 | 18 | 1 | 53
  Male | 10 | 11 | 6 | 16 | 11 | 2 | 56

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: During this follow-up study, it was planned to collect data from Year 16 through to Year 20 after primary vaccination. By the time the study protocol was approved, it was too late to collect data on Year 16. Therefore, the table presents mean concentrations expressed in milli-international units/milliliter (mIU/mL) at years 17, 18, 19 and 20.
Time Frame: Years 17, 18, 19 and 20.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBV 5 Group | HBV 2 Group | HBV 1 Group | HBV 4 Group | HBV 3 Group | HBV 6 Group
Number analyzed (Participants) | 17 | 20 | 17 | 23 | 29 | 3
mIU/mL
  Year 17 | 87.6 [27.6 to 278.2] | 43.8 [22.0 to 87.4] | 143.4 [39.2 to 523.9] | 34.4 [12.3 to 95.8] | 90.9 [45.8 to 180.3] | 10.6 [0.4 to 251.0]
  Year 18 | 96.2 [37.8 to 244.8] | 63.9 [32.2 to 126.6] | 121.6 [31.8 to 465.0] | 33.1 [15.2 to 72.2] | 89.1 [43.8 to 181.3] | 19.2 [0.0 to 2615400000]
  Year 19 | 37.4 [14.8 to 94.4] | 34.5 [20.6 to 57.7] | 108.1 [30.6 to 382.8] | 22.5 [11.7 to 43.6] | 62.1 [30.7 to 125.6] | 26.9 [2.0 to 363.6]
  Year 20 | 46.4 [19.6 to 109.8] | 25.8 [14.4 to 46.3] | 101.8 [28.7 to 361.7] | 20.3 [10.2 to 40.6] | 55.5 [30.1 to 102.1] | 12.8 [0.0 to 7642461]

2. Primary Outcome: Prevalence of Serological Markers for Hepatitis B Infection
Description: It was initially planned to collect data from Year 16 through to Year 20 after primary vaccination. By the time the study protocol was approved, it was too late to collect data on Year 16. Only the subjects positive for HBsAg or anti Hepatitis B core antigen (anti-HBc) were tested for HBeAg & anti-HBe
Time Frame: Years 17, 18, 19 and 20.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | HBV 5 Group | HBV 2 Group | HBV 1 Group | HBV 4 Group | HBV 3 Group | HBV 6 Group
Number analyzed (Participants) | 17 | 20 | 17 | 23 | 29 | 3
Percentage of participants (%)
  Year 17, HBsAg Negative | 100 | 93.7 | 100 | 100 | 96.3 | 100
  Year 17, HBsAg Positive | 0 | 6.3 | 0 | 0 | 3.7 | 0
  Year 17, Anti HBc Negative | 100 | 68.7 | 78.6 | 100 | 100 | 100
  Year 17, Anti HBc Positive | 0 | 31.3 | 21.4 | 0 | 0 | 0
  Year 17, HBeAg Negative | 0 | 100 | 100 | 0 | 100 | 0
  Year 17, HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0
  Year 17, Anti HBeAg Negative | 0 | 80 | 100 | 0 | 100 | 0
  Year 17, Anti HBeAg Positive | 0 | 20 | 0 | 0 | 0 | 0
  Year 18, HBsAg Negative | 100 | 100 | 100 | 100 | 96.4 | 100
  Year 18, HBsAg Positive | 0 | 0 | 0 | 0 | 3.6 | 0
  Year 18, Anti HBc Negative | 94.1 | 75 | 71.4 | 100 | 100 | 100
  Year 18, Anti HBc Positive | 5.9 | 25 | 28.6 | 0 | 0 | 0
  Year 18, HBeAg Negative | 100 | 100 | 100 | 0 | 100 | 0
  Year 18, HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0
  Year 18, Anti HBeAg Negative | 100 | 100 | 100 | 0 | 100 | 0
  Year 18, Anti HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0
  Year 19, HBsAg Negative | 92.9 | 94.1 | 100 | 85 | 82.1 | 75
  Year 19, HBsAg Positive | 7.1 | 5.9 | 0 | 15 | 17.9 | 25
  Year 19, Anti HBc Negative | 100 | 76.5 | 78.6 | 95 | 100 | 100
  Year 19, Anti HBc Positive | 0 | 23.5 | 21.4 | 5 | 0 | 0
  Year 19, HBeAg Negative | 100 | 100 | 100 | 100 | 80 | 100
  Year 19, HBeAg Positive | 0 | 0 | 0 | 0 | 20 | 0
  Year 19, Anti HBeAg Negative | 100 | 100 | 100 | 100 | 100 | 100
  Year 19, Anti HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0
  Year 20, HBsAg Negative | 100 | 76.5 | 92.9 | 78.9 | 84.6 | 100
  Year 20, HBsAg Positive | 0 | 23.5 | 7.1 | 21.1 | 15.4 | 0
  Year 20, Anti HBc Negative | 93.7 | 76.5 | 78.6 | 100 | 100 | 100
  Year 20, Anti HBc Positive | 6.3 | 23.5 | 21.4 | 0 | 0 | 0
  Year 20, HBeAg Negative | 100 | 100 | 100 | 100 | 100 | 0
  Year 20, HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0
  Year 20, Anti HBeAg Negative | 100 | 100 | 100 | 100 | 100 | 0
  Year 20, Anti HBeAg Positive | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Clinical Review for Hepatitis B Infection Status
Description: Chronic hepatitis B (HB) carrier is defined as positive for anti-HBc AND HBsAg at two or more consecutive time points
Time Frame: Over the entire 4 year follow up period (17 - 20 years)
Measure: Number; unit: participants
Arm/Group | HBV 5 Group | HBV 2 Group | HBV 1 Group | HBV 4 Group | HBV 3 Group | HBV 6 Group
Number analyzed (Participants) | 17 | 20 | 17 | 23 | 29 | 3
participants
  Chronic HB carriers | 0 | 1 | 1 | 0 | 0 | 0
  Chronic HB carriers among primary study responders | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.